CLINICAL TRIAL: NCT02126137
Title: A Pilot Study of the Effect of Ezetimibe in Patients With Chronic Hepatitis C Infection
Brief Title: Pilot Study of Ezetimibe for Chronic Hepatitis C Virus (HCV) Infection
Acronym: EZE-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-199; 1130357 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Ezetimibe; Cholesterol; Host
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ezetimibe (Experimental): Ezetimibe administered by mouth 10 mg BID for 12 weeks
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe

SUMMARY:
Infection by hepatitis C virus (HCV) affects more than 170 million people in the World and 80.000 in Chile. It causes more deaths than HIV infection in the US and is a leading cause for liver transplantation in Chile. Even though treatments are evolving with new direct antiviral agents (DAAs) that are increasing response rates, there are several issues with these new approaches, including increased toxicity, need for using interferon and ribavirin, complex algorithms of treatment, high cost, limited effectivity in certain groups (liver transplant patients) and drug interactions. Treatments targeted at host factors required for the viral cycle are becoming increasingly explored as an alternative or complement to DAAs. It has been recently described that Niemann-Pick C1-like 1 (NPC1L1), the intestinal receptor of cholesterol, serves as an entry factor for HCV. NPC1L1 is, therefore, a key transporter in the enterohepatic cycle of cholesterol. NPC1L1 can be blocked with ezetimibe, which is an approved and generally safe drug used for the management of hypercholesterolemia. Our hypothesis posits that blocking HCV entry to the hepatocyte or intestinal HCV reabsorption with ezetimibe may have an antiviral effect. In the study, we will administer ezetimibe 20 mg/d to 20 patients with stable chronic hepatitis C for 12 weeks and assess changes in HCV RNA and core antigen in plasma, bile and feces.

ELIGIBILITY:
Inclusion criteria:

* Chronic hepatitis C defined as detectable HCV RNA for more than 6 months.
* Age > 18 years old.
* Compensated liver disease (bilirubin < 3mg/dL, unless having Gilbert´s syndrome, albumin > 3 g/dL, INR < 2, no hepatic encephalopathy, no ascites or recent -1 month- history of variceal bleeding).
* HCV RNA level > 10.000 IU/mL.
* Signed informed consent document.

Exclusion criteria:

* History of cholecystectomy or known gallstones.
* Current HCV antiviral treatment.
* Medications for dyslipidemia in the preceding 2 months.
* Abdominal surgery that could alter biliary or intestinal anatomy.
* Evidence of sitosterolemia.
* Negative pregnancy test in urine (for females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
HCV plasma viral load | 12 weeks

SECONDARY OUTCOMES:
HCV biliary viral load | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Soza, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Department of Gastroenterology, Pontificia Universidad Católica de Chile, Santiago, Metropolitan, Chile

REFERENCES:
- [Background] Sainz B Jr, Barretto N, Martin DN, Hiraga N, Imamura M, Hussain S, Marsh KA, Yu X, Chayama K, Alrefai WA, Uprichard SL. Identification of the Niemann-Pick C1-like 1 cholesterol absorption receptor as a new hepatitis C virus entry factor. Nat Med. 2012 Jan 8;18(2):281-5. doi: 10.1038/nm.2581. PMID 22231557
- See also: Centro de Investigación Clínica UC (CICUC) — http://medicina.uc.cl/CICUC-centro-investigacion-clinica
- See also: Information related to hepatitis C / Información de hepatitis por virus C (Spanish) — http://hepatitis.cl